CLINICAL TRIAL: NCT03270995
Title: Efficacy of a Cognitive-existential Intervention to Address Fear of Recurrence in Women With Cancer: a Randomized Controlled Clinical Trial
Brief Title: Cognitive-Existential Group Therapy to Reduce Fear of Cancer Recurrence: A RCT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Princess Margaret Hospital, Canada (Other); University of Ottawa (Other); Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Christine Maheu, Principal Investigator, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT FCR
Record Dates: First submitted 2016-03-17; First posted 2017-09-01 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms
Keywords: breast cancer; gynecological cancer; fear of cancer recurrence; clinical trial; randomized controlled trial; group therapy; intervention; cognitive-existential
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Behavioral:Cognitive Existential Therapy Group 1- Weekly two-hour group sessions
  Interventions: Behavioral: Cognitive Existential Therapy Group 1
- Group 2 (Active Comparator): Behavioral: Supportive Therapy Group 2- Weekly two-hour group sessions
  Interventions: Behavioral: Supportive Therapy Group 2

INTERVENTIONS:
Behavioral: Cognitive Existential Therapy Group 1 — Six group sessions of two hour each using a cognitive-existential group approach
  Arms: Group 1
Behavioral: Supportive Therapy Group 2 — Six group session of two hour each using a supportive group approach.
  Arms: Group 2

SUMMARY:
Studies show that cancer survivors have unmet needs, the most frequently cited being fear of recurrence (FCR). Moderate to high levels of FCR have been reported by as much as 49% of cancer patients and are more prevalent among women. FCR is associated with psychological distress, lower quality of life, and increased health care utilization. Little evidence exists that these problems are being addressed by current medical management.

DETAILED DESCRIPTION:
The present study aims to further test this cognitive-existential group intervention for FCR in a randomized control clinical trial with women with breast or gynecological cancer. Participants will be recruited from Princess Margaret Hospital, Mount Sinai Hospital, the Jewish General Hospital, and the Ottawa Hospital. 144 cancer patients will be randomized to either receive the 6 week cognitive-existential group intervention or to a control group. The control group will also consist of six weekly sessions during which participants will discuss the challenges of living with a cancer diagnosis, but without a clear focus on FCR. Women randomized to participate in the study will a) be 18 years or older; b) have a first diagnosis of breast or gynecological cancer with stages between IIII; c) be disease free at the start of the group; d) gave clinical levels of fear of cancer recurrence; e) have clinical levels of distress; and f) have completed their cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. first diagnosis of BC or GC with stages between I-III;
2. disease-free at the start of the group;
3. women aged 18 years or older;
4. completion of treatment, with the exception of adjuvant chemotherapy or hormonal replacement therapy

Exclusion Criteria:

1. non-English speakers
2. previous cancer recurrence
3. enrolled in another group psychotherapy at the time of the start of the study or during the course of the 6 sessions
4. unresolved mental health disorder judged to be clinically contra-indicated and/or likely to affect the group work, based on disclosure by the potential participant or clinically identified by the group leader.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-10; Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Fear of cancer recurrence inventory | up to 12 months post-intervention follow-up
  Fear of cancer recurrence will be measured using the Fear of Cancer Recurrence Inventory (FCRI). The FCRI is a 42-item questionnaire that includes a global score as well as seven sub-scales including triggers, severity, psychological distress, functional impairment, insight, reassurance, and coping strategies. A score of 13 or greater on the nine-item severity subscale (range 0-36) indicates clinical level of FCR [55]. The instrument has been shown to have adequate reliability and validity (construct validity; r=0.68 to 0.77; and reliability scores; α=0.95).

SECONDARY OUTCOMES:
Cancer-specific distress | Pre- two weeks prior to the intervention, Post-one week after the end of the intervention, and three (T3) and six months (T4) following the end of the intervention
  Cancer-specific distress with the Impact of Event Scale (IES)]; The IES is a 15 items questionnaires that assesses cancer distress. It has two sub-scales, intrusive thoughts and avoidance, which provide a total score.
Perceived risk of cancer recurrence | Pre- two weeks prior to the intervention, Post-one week after the end of the intervention, and three (T3) and six months (T4) following the end of the intervention
  Perceived risk of cancer recurrence will be assessed using a one-item question where respondents indicate their level of perceived personal risk for a cancer recurrence over the last two days.
Intolerance of uncertainty | Pre- two weeks prior to the intervention, Post-one week after the end of the intervention, and three (T3) and six months (T4) following the end of the intervention
  Intolerance of uncertainty with be measured with the Intolerance of Uncertainty Scale (IUS) [58]. The IUS is a 27-item four-factor questionnaire that represents uncertainty as stressful and upsetting, uncertainty as leading to the inability to act, uncertain events as being negative and to be avoided, and being uncertain as unfair.
Uncertainty in Illness | Pre- two weeks prior to the intervention, Post-one week after the end of the intervention, and three (T3) and six months (T4) following the end of the intervention
  Uncertainty in Illness will be measured by the Mishel Uncertainty in Illness Scale (MUIS-C) [59]. The MUIS-C consists of 23 items rated on a five-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Maheu, RN, PhD, Principal Investigator — McGill University and University Health Network
Locations (3):
- Canada (3):
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maheu C, Lebel S, Courbasson C, Lefebvre M, Singh M, Bernstein LJ, Muraca L, Benea A, Jolicoeur L, Harris C, Ramanakumar AV, Ferguson S, Sidani S. Protocol of a randomized controlled trial of the fear of recurrence therapy (FORT) intervention for women with breast or gynecological cancer. BMC Cancer. 2016 Apr 25;16:291. doi: 10.1186/s12885-016-2326-x. PMID 27112319
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27112319